CLINICAL TRIAL: NCT04910542
Title: Epidemiologic Intelligence Network (EpI-Net) to Promote COVID-19 Testing and Prevention Practices Among Socially Vulnerable Communities in Puerto Rico
Brief Title: Epidemiologic Intelligence Network (EpI-Net) to Promote COVID-19 Testing
Acronym: EpI-Net
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce Medical School Foundation, Inc. (Industry)
Collaborators: Duke University (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3R21MD013674-02S2 (NIH)
Record Dates: First submitted 2021-03-30; First posted 2021-06-02 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study employs a mixed-methods design for intervention trials. This method is appropriate for epidemiological interventions framed under community engagement practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EpI-Net community intervention (Other): The Epidemiological Intelligence Network Intervention (Epi-Net) is a group of field epidemiology tools for test, trace and isolate using a community-based approach. The overall goal of Epi-Net is to increase uptake of COVID-19 testing and prevention practices among socially vulnerable communities in Puerto Rico. The intervention intends to impact COVID-19 risk perception, decrease COVID-19 testing barriers, increase testing uptake and increase health promotion strategies.
  Interventions: Other: Epi-Net Intervention

INTERVENTIONS:
Other: Epi-Net Intervention — The Epidemiological Intelligence Network Intervention (Epi-Net) is a group of field epidemiology tools for test, trace and isolate using a community-based approach. The overall goal of Epi-Net is to increase uptake of COVID-19 testing and prevention practices among socially vulnerable communities in Puerto Rico. The intervention intends to impact COVID-19 risk perception, decrease COVID-19 testing barriers, increase testing uptake and increase health promotion strategies.

SUMMARY:
The investigators propose a mixed-methods intervention design to evaluate the acceptability of epidemic intelligence (EpI-Net) intervention using Community Engagement (CE) principles to promote COVID-19 testing and prevention practices in socially vulnerable communities in PR. The team hypothesizes that the integration of lay community leaders, trained in the use of COVID-19 prevention technology tools (EpI-Net), will result in increased COVID-19 testing uptake and prevention practices among the targeted socially and epidemiologically vulnerable communities in Puerto Rico.

DETAILED DESCRIPTION:
On March 11, 2020, the World Health Organization (WHO) officially declared the SARS-CoV-2 (COVID-19) outbreak a pandemic. In Puerto Rico (PR), the first COVID-19 case was confirmed early March 2020. To date, cases have exponentially increased partly due to the lifting of locked-down restriction by the PR government, limited COVID-19 testing, and contact tracing. As a major Public Health Emergency (PHE), the COVID-19 pandemic has disproportionally affected racial and ethnic minorities as well as patients with chronic health conditions. Specifically, residents of PR are socially and epidemiologically vulnerable with one of the highest prevalence rates for chronic diseases (diabetes, hypertension, obesity, HIV) prevalence rates and arbovirus-related diseases, such as Zika and Dengue. Puerto Ricans living on the island are also particularly vulnerable to the current overlapping of the COVID-19 pandemic and natural disasters (earthquake, hurricanes/storms). Limited access to molecular COVID-19 testing throughout PR has been a significant challenge. Without adequate testing, estimates for SARS-CoV-2 (COVID-19) infection rates are limited, and targeted prevention efforts (focused testing) be inadequate. Ponce Research Institute (PRI) with the support of Ponce Health Sciences University (PHSU) - leads the COVID-19 outreach efforts in PR related to earthquake aftershocks, tropical storms, and the COVID-19 pandemic. The PHSU-PRI Research Center for Minority Institutions-Community Engagement Core (RCMI-CEC) leaders in collaboration with community leaders, implemented the COVID-19 prevention education initiative which targets socially vulnerable populations in southern Puerto Rico (the earthquake and aftershocks epicenter). Also, PHSU-PRI epidemiologists (led by Dr. Marzán-Rodríguez, MPI) developed a web-based COVID-19 Epidemiologic Surveillance System (ESSS) in collaboration with the Puerto Rico Public Health Trust (PRPHT, a community partner for this grant) with more than 46,000 surveys completed up to September 2020. The ESSS tool is an online geocoded survey that identifies real-time COVID-19-related symptoms during the last 24 hours; and thus, prioritizes communities for COVID-19 testing. The ESSS tool can be easily accessed on the PRPHT website. Leveraging the current PHSU-PRI COVID-19 prevention efforts and the ESSS infrastructure, the research team proposes a mixed-methods approach for intervention trials for dissecting the impact of an epidemic intelligence (EpI-Net) community-based intervention aimed at increasing COVID-19 testing uptake and prevention practices among socially vulnerable communities in PR. Under Aim 1, the team will train lay community leaders on the use and application of COVID-19 early detection epidemic intelligence tools. Under Aim 2, the team will identify and understand the individual (beliefs and behaviors), social, cultural, and contextual factors facilitating the adoption and adherence to routine COVID-19 testing and prevention practices. Under Aim 3, the team will test EpI-Net intervention preliminary impact on increasing COVID-19 testing uptake and prevention practices among socially vulnerable communities in PR. The working hypothesis is that the integration of lay community leaders, trained in the use of COVID-19 prevention technology tools (EpI-Net), will result in increased COVID-19 testing uptake and prevention practices among the targeted socially and epidemiolocal vulnerable communities in Puerto Rico.

ELIGIBILITY:
Inclusion Criteria:

* Community Leaders Eligibility Criteria: After the team's identified the community, with the support of the community partners and the Community Scientific Advisory Committee, we will invite community leaders to be part of the EpI-Net training. The inclusion criteria for the community leaders to be trained in EpI-Net activities are: (1) >21 years of age, (2) living in a socially vulnerable community for COVID-19 according to the CDC-SVI; (3) self-identified as a Latino/Hispanic and; (4) be able to provide support for the EpI- Net implementation process in their communities.
* In-depth Interview Participants' Eligibility Criteria: The eligibility criteria for the qualitative interviews will be: (1) >21 years old, (2) living in a socially vulnerable community for COVID-19 according to the CDC-SVI (Ref); (3) self-identified as a Latino/Hispanic; (4) be part of the participant municipalities at the RCMI-CEC program or PRPHT network and (5) be able to complete an interview.
* Communities' Eligibility Criteria: Based on factors associated with COVID-19 complications such as high chronic disease prevalence (including obesity rates), age group distribution, population density and socioeconomic status, and COVID-19 positivity rates, we will preliminarily identify potential municipalities to be impacted by this project.Those preliminar municipalities are: Ponce, Guánica, Vieques, San Juan, Loíza, Vega Alta, Aibonito, Yauco, Mayagüez and Naranjito. Once municipalities are identified, the team will rely on the CDC-SVI index to identify the communities (within these municipalities) with higher socially vulnerability.
* Community Survey Eligibility Criteria: The eligibility criteria for the community survey will be: (1) >21 years old, (2) living in a socially vulnerable community for COVID-19 according to the CDC-SVI (Ref); (3) self-identified as a Latino/Hispanic; (4) be part of the participant municipalities at the RCMI-CEC program or PRPHT network and (5) be able to complete an interview.
* Epidemiological Syndromic Surveillance System (ESSS) Eligibility Criteria: Participants eligible to complete the ESSS are residents of Puerto Rico, 18 years of age and older.

Exclusion Criteria:

* Children and adolescents are excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3301 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change COVID-19 testing uptake | Five months per community
  By June 2022, EpI-Net intervention will have provided 2,700 COVID-19 RT-PCR tests among six socially vulnerable communities in PR.
  1. Tabulation of PCR tests by test ID and date of sample collection.
  2. Tabulation of PCR test results received by the molecular laboratory.
  i.COVID-19 test results by EpI-NET uploaded to REDCap servers. c.TESTING ASSESSMENT i.% of participants who received a COVID-19 RT-PCR tests for the first time.
  1. Have you ever been tested for COVID-19?
     1. No
     2. Yes
     3. Prefer not to answer
  2. How did you get tested for your most recent test?
     1. Nasal Swab (Antigen)
     2. Swab in the nose and throat (PCR)
     3. Blood
     4. Saliva

SECONDARY OUTCOMES:
Change Covid-19 positivity rates <5% | Five months per community
  Assessment
  a.Baseline COVID-19 positivity rate vs 5 months COVID-19 positivity rate. i.Have you ever tested positive for COVID-19?/Yes;/No/I don't know/Prefer not to answer ii.In which month did you first test positive for COVID-19?/January/February/March/ April/May/June/July;/August;/September/October/November/December iii.In what year did you first test positive for COVID-19? /2019/2020/2021 iv.In what month did you have your most recent COVID-19 test?/January/February/March/ April/May/June/July;/August;/September/October/November/December v.What year was the most recent COVID-19 test done?/2019/2020/2021 vi.What was the result of your most recent COVID-19 test?/Negative/Positive/I never obtained the results/Undetermined/I don't know/Prefer not to answer
Covid-19 prevention practices awareness of >25% | Five months per community
  Assessment
  a.Baseline COVID-19 prevention practices awareness vs 5 months COVID-19 prevention practices awareness i.What messages have you heard in your VV about preventing the spread of COVID-19?/Wear a protective face cover/Disinfect different surfaces/Wash hands frequently with soap and water/Avoid group meetings/Disinfect packages, boxes, or mail/Disinfect grocery bags or packages/Wash fruits, vegetables and other food products with bleach/Take medications/Take vitamins or essential oils/Do not travel abroad/Do not travel within the island/Other/I have not heard any messages/Don't know/Prefer not to answer ii.Currently,how worried are you or the members of your VV by the contagion of COVID-19? /Very/Somewhat/Not prepared at all/Don't know/Prefer not to answer iii.How prepared was your VV for the COVID-19 pandemic and related stay-at-home orders?/Very/Somewhat/Not prepared at all/Don't know/Prefer not to answer
Covid-19 prevention practices uptake of >25% | Five months per community
  Assessment Baseline COVID-19 prevention practices uptake vs 5 months COVID-19 prevention practices uptake.
  i.Someone who has completed quarantine does not pose a risk of infection to the public or to themselves ii.Do you or a member of your VV think you had COVID-19 but were never tested? In response to the COVID-19 pandemic are you or members of your VV; iii. currently wearing a mask in public places? iv.currently avoiding meetings? v.currently conduct food washing (eg, bags)? vi.currently do vegetable washing? vii.currently wear gloves in public? viii.currently have hand disinfectant if you can't wash your hands? ix. In the past 30 days how often have you and the members of your VV left your home? In the past 30 days have you or members of your VV visited; x.a Beauty salon, massage center? xi.a Public park or beach? xii.the Interior of the restaurant? xiii.an Open-air restaurant? xiv.a Doctor's office?

CONTACTS AND LOCATIONS:
Overall Officials: Eida M Castro, PsyD, Principal Investigator — Ponce Medical School Foundation
Locations (1):
- Ponce Medical School Foundation, Ponce, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
At this moment, no individual personal data will be available to others researchers

REFERENCES:
- [Derived] Marzan-Rodriguez M, Muniz-Rodriguez K, Morales LM, Martinez IS, Torres-Borrero N, Castro-Figueroa EM. Epidemiological intelligence community network intervention: a community response for COVID-19 community transmission. BMC Public Health. 2023 Jun 1;23(1):1044. doi: 10.1186/s12889-023-15727-3. PMID 37264399